CLINICAL TRIAL: NCT00200681
Title: Etude Multicentrique Ouverte Randomisée de Phase III Comparant l'Association de VELCADE®-Dexaméthasone à la Chimiothérapie de Type VAD Pour le Traitement Des Patients Porteurs de Myélome Multiple de Novo Jusqu'à l'âge de 65 Ans
Brief Title: IFM 2005-01: Velcade/Dexamethasone Versus Vincristine/Adriamycin (Doxorubicin)/Dexamethasone (VAD) for the Treatment of Patients With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: BRD 04/11-J
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Multiple Myeloma
Keywords: Secretory Multiple Myeloma; First line treatment; Velcade®; autograft; Newly diagnosed secretory Multiple Myeloma (MM)
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Velcade

SUMMARY:
This is an open-label, multi-centre, randomised Phase III study, looking at a series of 480 patients up to the age of 65 with newly diagnosed multiple myeloma (MM) not previously treated. They will receive VAD or Velcade®/dexamethasone combination as induction treatment plus/minus (±) dexamethasone/cyclophosphamide/etoposide/cisplatin (DCEP) followed by autograft as first-line therapy, as the investigators try to compare the complete remission (CR) rate (with negative or positive immunofixation) at the end of their induction treatment.

DETAILED DESCRIPTION:
After their written informed consent has been obtained and their eligibility verified, patients are randomised between 4 treatment arms: A1 VAD (4 cycles); A2 VAD (4 cycles) followed by DCEP (2 cycles); B1 Velcade® + dexamethasone (4 cycles); B2 Velcade® + dexamethasone (4 cycles) followed by DCEP (2 cycles) A1, A2, B1, B2 + autograft. Randomisation will be stratified on the basis of the initial b2 microglobulin level (> or < 3 mg/l) and the presence of chromosome 13 abnormalities identified by FISH analysis. VAD: Vincristine/Adriamycin/Dexamethasone; DCEP: Dexamethasone/Cyclophosphamide/ Etoposide/Cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed MM according to the criteria of the South West Oncology Group (SWOG)
* Not previously treated, apart from local radiotherapy, in the case of a threatening or incapacitating lesion, and/or a 4-day block of dexamethasone (40 mg/mL) in an emergency
* Stage II or III disease according to the Durie and Salmon classification or Stage I disease with symptomatic bone lesion
* < 65 years of age
* Ability to give signed informed consent
* Secretion of a measurable monoclonal spike (> 10 g/l in the serum or 0.2 g/24h in the urine)
* Negative pregnancy test at inclusion (if necessary)
* Absence of active infection. In the case of infection, appropriate antibiotic therapy must be administered and patients must have been apyretic for 48 hours before the start of treatment with VAD or Velcade®/dexamethasone

Exclusion Criteria:

* ECOG performance status > 2
* History of cancer (other than basal cell carcinoma or carcinoma of the cervix in situ)
* Life expectancy < 2 months
* Confirmed amyloidosis
* Positive HIV serology
* Serious psychiatric item in the history
* Renal failure requiring dialysis
* Uncontrolled diabetes, contra-indicating the use of corticosteroids
* Peripheral neuropathy National Cancer Institute (NCI) grade > 2 (Annex 5)
* Clinical signs of heart failure or coronary heart disease
* Bilirubin > 3 x normal
* Transaminases or gamma-glutamyl transpeptidase (GT) > 4 x normal
* Platelets < 50 x 10^9/l during the 15 days prior to inclusion
* Neutrophils < 0.75 x 10^9/l during the 15 days prior to inclusion
* Use of an investigational medicinal product during the 30 days prior to inclusion
* Known hypersensitivity to bortezomib, boron or mannitol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2005-06; Primary Completion 2008-01 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To compare the CR rate (with negative or positive immunofixation) obtained with VAD or the Velcade®/dexamethasone combination used as induction treatment in patients up to the age of 65 with newly diagnosed MM, at the end of this induction treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Harousseau, MD PHD, Principal Investigator — Intergroupe Francophone du Myélome (IFM)
Locations (1):
- CHU de Nantes, Service d'Hématologie, Nantes, France

REFERENCES:
- [Derived] Sonneveld P, Goldschmidt H, Rosinol L, Blade J, Lahuerta JJ, Cavo M, Tacchetti P, Zamagni E, Attal M, Lokhorst HM, Desai A, Cakana A, Liu K, van de Velde H, Esseltine DL, Moreau P. Bortezomib-based versus nonbortezomib-based induction treatment before autologous stem-cell transplantation in patients with previously untreated multiple myeloma: a meta-analysis of phase III randomized, controlled trials. J Clin Oncol. 2013 Sep 10;31(26):3279-87. doi: 10.1200/JCO.2012.48.4626. Epub 2013 Jul 29. PMID 23897961
- [Derived] Corthals SL, Kuiper R, Johnson DC, Sonneveld P, Hajek R, van der Holt B, Magrangeas F, Goldschmidt H, Morgan GJ, Avet-Loiseau H. Genetic factors underlying the risk of bortezomib induced peripheral neuropathy in multiple myeloma patients. Haematologica. 2011 Nov;96(11):1728-32. doi: 10.3324/haematol.2011.041434. Epub 2011 Jul 26. PMID 21791469
- [Derived] Moreau P, Attal M, Pegourie B, Planche L, Hulin C, Facon T, Stoppa AM, Fuzibet JG, Grosbois B, Doyen C, Ketterer N, Sebban C, Kolb B, Chaleteix C, Dib M, Voillat L, Fontan J, Garderet L, Jaubert J, Mathiot C, Esseltine D, Avet-Loiseau H, Harousseau JL; IFM 2005-01 study investigators. Achievement of VGPR to induction therapy is an important prognostic factor for longer PFS in the IFM 2005-01 trial. Blood. 2011 Mar 17;117(11):3041-4. doi: 10.1182/blood-2010-08-300863. Epub 2010 Nov 23. PMID 21098740